CLINICAL TRIAL: NCT03015675
Title: Phase Ⅲ Study of IV Ascorbic Acid in Combination With XELOX vs Treatment With XELOX Alone as First-line Therapy for Advanced Gastric Cancer
Brief Title: IV Ascorbic Acid in Advanced Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCV 001
Record Dates: First submitted 2017-01-08; First posted 2017-01-10 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Ascorbic Acid; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ascorbic Acid with mFOLFOX6 group (Experimental): Ascorbic Acid with mFOLFOX6 Ascorbic Acid (20g/day, D1-3) every 2 weeks
  mFOLOX6:
  * Oxaliplatin 85 mg/m² d1 concurrent with
  * Leucovorin 400 mg/m², followed by
  * Bolus 5FU 400 mg/m² , followed by
  * Infusional 5FU 2400 mg/m² over 46 hours, every 2 weeks
  Interventions: Drug: ascorbic acid; Drug: mFOLFOX6
- mFOLFOX6 group (Active Comparator): mFOLOX6:
  * Oxaliplatin 85 mg/m² d1 concurrent with
  * Leucovorin 400 mg/m², followed by
  * Bolus 5FU 400 mg/m² , followed by
  * Infusional 5FU 2400 mg/m² over 46 hours, every 2 weeks
  Interventions: Drug: mFOLFOX6

INTERVENTIONS:
Drug: ascorbic acid — 20g/day, D1-3, every 2 weeks
  Other Names: vitamin C
  Arms: Ascorbic Acid with mFOLFOX6 group
Drug: mFOLFOX6 — mFOLFOX6
  * Oxaliplatin 85 mg/m² d1 concurrent with
  * Leucovorin 400 mg/m², followed by
  * Bolus 5FU 400 mg/m² , followed by
  * Infusional 5FU 2400 mg/m² over 46 hours, every 2 weeks
  Other Names: chemotherapy

SUMMARY:
Linus Pauling and Dr Ewan Cameron have published two retrospective studies about using high dose vitamin C to treat cancer patients forty years ago. Their studies have shown that high dose vitamin C usage could significantly prolong overall survival of patients with advanced cancer. Recently, preclinical study has shown that human colorectal cancer cells harboring KRAS or BRAF mutations are selectively killed by high levels of ascorbic acid (AA). High dose of AA impairs tumor growth in Apc/KRASG12D mutant mice. Previous phaseⅠclinical trials have found that high dose (1.5g/kg or 90g/m2) iv AA is well tolerated in cancer patients. This protocol is a phase Ⅲ, study of ascorbic acid (AA) infusions combined with treatment with mFOLOX6 versus mFOLOX6 alone as first-line therapy in patients with recurrent or advanced gastric cancer.

DETAILED DESCRIPTION:
Linus Pauling and Dr Ewan Cameron have published two retrospective studies about using high dose vitamin C to treat cancer patients forty years ago. Their studies have shown that high dose vitamin C usage could significantly prolong overall survival of patients with advanced cancer. Recently, preclinical study has shown that human colorectal cancer cells harboring KRAS or BRAF mutations are selectively killed by high levels of ascorbic acid (AA). High dose of AA impairs tumor growth in Apc/KRASG12D mutant mice. Previous phaseⅠclinical trials have found that high dose (1.5g/kg or 90g/m2) iv AA is well tolerated in cancer patients. This protocol is a phase Ⅲ, study of ascorbic acid (AA) infusions combined with treatment with mFOLOX6 versus mFOLOX6 alone as first-line therapy in patients with recurrent or advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

Age≥18 years, ≤75 years; Histologically proven metastatic adenocarcinoma of stomach (stage 4 disease), unresectable metastatic disease; G6PD status > lower limit of normal; Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2; Life expectancy of at least 12 weeks; ANC ≥1,500/mm3; Hemoglobin > 8g/dL; platelet ≥ 100,000/mm3; Laboratory at baseline evaluation for inclusion in the study: creatinine ≤1.5X upper limit [if the creatinine is elevated, but ≤1.5X the ULN, a 24 hour ;creatinine clearance will be obtained, Creatinine clearance > 50 mL/min (calculated according to Cockroft and Gault)]; Transaminase (AST/ALT) ≤2.5X upper limit of normal and bilirubin levels ≤1.5X upper limit of normal without liver metastasis; Transaminase (AST/ALT) ≤5X upper limit of normal and bilirubin levels ≤1.5X upper limit of normal with liver metastasis; Women of childbearing potential will confirm a negative pregnancy test and must practice effective contraception during the study; Written informed consent

Exclusion Criteria:

Prior treatment for metastatic disease (adjuvant therapy with fluoropyrimidines +/-oxaliplatin based regimens allowed if stopped 12 months prior to registration on study); Surgery (excluding diagnostic biopsy) or irradiation within 3 weeks prior to study entry; Administration of any investigational drug or agent/procedure, i.e. participation in another trial within 4 weeks before beginning treatment; Concurrent chronic systemic immune therapy, chemotherapy, radiation therapy (palliative radiation therapy allowed) or hormone therapy not indicated in the study protocol; Brain metastasis (known or suspected); Pregnant or lactating women; Other uncontrolled concomitant illness, including serious uncontrolled intercurrent infection; Known allergy or any other adverse reaction to any of the drugs or to any related compound; Previous (within 5 years) or concurrent malignancies at other sites with the exception of surgically cured or adequately treated carcinoma in-situ of the cervix and basal cell carcinoma of the skin; Patients who are on strong inducers of CYP3A4 which include but are not limited to: Aminoglutethimide, Bexarotene, Bosentan, Carbamazepine, Dexamethasone, Efavirenz, Fosphenytoin, Griseofulvin, Modafinil, Nafcillin, Nevirapine, Oxcarbazepine, Phenobarbital, Phenytoin, Primidone, Rifabutin, Rifampin, Rifapentine, St. John's wort; Medical, social or psychological condition which, in the opinion of the investigator, would not permit the patient to complete the study or sign meaningful informed consent; Organ allograft requiring immunosuppressive therapy; Patients with HIV infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-03-12 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | up to 5 years
  Time-to-event outcome measure (initial disease progression) measured in days from cycle 1 day 1 to day of first progression as defined by RECIST1.1 criteria from NCI

SECONDARY OUTCOMES:
Overall Survival | up to 5 years
  Time to event outcome measure (death), measured in days from cycle 1 day 1
Response Rate | up to 5 years
  To utilize CT or PET/CT scans to assess overall tumor response rate (complete and partial response) and evaluate disease progression in subjects with advanced or recurrent RAS mutant colorectal cancer treated with the combination of ascorbic acid and FOLOX/FORFIRI +/- bevacizumab versus treatment with FOLFOX/FORFIRI +/- bevacizumab alone

CONTACTS AND LOCATIONS:
Overall Officials: Rui-hua Xu, MD.,PhD., Principal Investigator — Sun Yat-sen University
Locations (1):
- Medical Oncology,Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided